CLINICAL TRIAL: NCT02240485
Title: Integrative Couple Treatment for Pathological Gambling or Individual Treatment: A Comparison of Efficacy
Brief Title: Integrative Couple Treatment for Pathological Gambling
Acronym: ICT-PG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université du Québec à Trois-Rivières (Other)
Responsible Party: Principal Investigator, Joël Tremblay, Principal Investigator, Université du Québec à Trois-Rivières
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CER-10-156-06.13
Record Dates: First submitted 2014-08-04; First posted 2014-09-15 (Estimated); Results first posted 2022-03-18 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Pathological Gambling
Keywords: Pathological gambling; Treatment; Marital relationship
MeSH Terms: conditions — Gambling | interventions — Couples Therapy; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrative Couple Treatment for Pathological Gambling (ICT-PG) (Experimental): Couple therapy: The experimental couple treatment is offered over 8 to 12 sessions of 90 minutes. The couple treatment called (Integrative Couple Treatment for Pathological Gambling - ICT-PG) is inspired by the "Alcohol Behavior Couple Therapy" from Epstein and McCrady, to which the team added diverse components to adjust to gamblers. During the sessions, the focus is on a) reducing/stopping gambling behaviors, b) helping the partner to stop behaviors facilitating gambling habits and rise the frequency of behaviors incompatible with gambling habits and c) improve marital components (communication, sharing positive moments, negotiation, mutual support).
  Interventions: Behavioral: Integrative Couple Treatment for Pathological Gambling (ICT-PG)
- Usual individual/group treatment (Active Comparator): Usual individual/group treatment: The control group receive individual or group treatment as already offered by the specialized centers in addiction.Their partner can receive individual intervention if desired.
  Interventions: Behavioral: Usual individual/group treatment

INTERVENTIONS:
Behavioral: Integrative Couple Treatment for Pathological Gambling (ICT-PG) — The experimental couple treatment is offered over 8 to 12 sessions of 90 minutes. The couple treatment called (Integrative Couple Therapy for Pathological Gambling - ICT-PG) is inspired by the "Alcohol Behavior Couple Therapy" from Epstein and McCrady, to which the team added diverse components to adjust to gamblers. During the sessions, the focus is on a) reducing/stopping gambling behaviors, b) helping the partner to stop behaviors facilitating gambling habits and rise the frequency of behaviors incompatible with gambling habits and c) improve marital components (communication, sharing positive moments, negotiation, mutual support).
  Other Names: Couple therapy
  Arms: Integrative Couple Treatment for Pathological Gambling (ICT-PG)
Behavioral: Usual individual/group treatment — The control group receive individual or group treatment as already offered by the specialized centers in addiction.Their partner can receive individual intervention if desired.
  Other Names: treatment as usual
  Arms: Usual individual/group treatment

SUMMARY:
The aim of the study is to compare marital treatment to individual treatment for pathological gambling.

DETAILED DESCRIPTION:
The study as two goals: evaluate the efficacy of couple treatment for pathological gambling and develop a better understanding of the individual (substance use, mental health) and couple dimensions (communication, marital satisfaction, violence) as intermediate variables explaining this efficacy. Couples will be randomized between the couple treatment and the treatment as usual (individual or group). The experimental couple treatment is offered over 8 to 12 sessions of 90 minutes. The couple treatment called (Integrative Couple Therapy for Pathological Gambling - ICT-PG) is inspired by the "Alcohol Behavior Couple Therapy" from Epstein and McCrady, to which the team added diverse components to adjust to gamblers. During the sessions, the focus is on a) reducing/stopping gambling behaviors, b) helping the partner to stop behaviors facilitating gambling habits and rise the frequency of behaviors incompatible with gambling habits and c) improve marital components (communication, sharing positive moments, negotiation, mutual support).

The control group receives individual or group treatment as already offered by the specialized centers in addiction. Their partner can receive individual intervention if desired. All participants are recruited in Specialized Addiction Treatment Centers in Quebec province, Canada. Evaluation of participants is done at admission, three, nine and 18 months post-admission.

Repeated measures ANOVA will be used to compared evolutions of groups over time. Multiple regression will allow the estimation of components roles into as intermediate variables to predict rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Living together for at least 1 year
* Diagnosis of pathological gambling (WMH-CIDI) during the last 12 months
* The gambler has not received treatment for their gambling for at least 6 months (excluding GA)
* Presence of gambling behavior in the past 3 months
* Degree of commitment to the couple indicating a desire to continue the relationship (score of 7 - MSI)

Exclusion Criteria:

* Alcohol/Drug Dependence gambler/partner (Severity of Alcohol Dependence Data questionnaire - SADD >17 included in DEBA-A; Severity of Dependence Scale - SDS > 5 Included in DEBA-D)
* Gambling problem for the partner (DEBA-Jeu > 10)
* Presence of serious acts of violence endangering the safety of both spouses (CTS-2)
* Disorder and serious mental health unstabilized one of two members of the couple (ASI: psychological scale)
* Antisocial personality disorder or severe limit ( GAIN: 9 + Scale BCS / CDS)
* Scenario with strong suicidal ideation or attempt in the last 30 days or less in the partner (ASI: psychological scale)
* Low degree of commitment in the relationship of a risk of separation (8 + MSI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-03-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joël Tremblay, Principal Investigator — Université du Québec à Trois-Rivières
Locations (1):
- Université du Québec à Trois-Rivières, Québec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tremblay J, Dufour M, Bertrand K, Saint-Jacques M, Ferland F, Blanchette-Martin N, Savard AC, Cote M, Berbiche D, Beaulieu M. Efficacy of a randomized controlled trial of integrative couple treatment for pathological gambling (ICT-PG): 10-month follow-up. J Consult Clin Psychol. 2023 Apr;91(4):221-233. doi: 10.1037/ccp0000765. Epub 2022 Dec 15. PMID 36521131

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was carried out in two phases:
  Phase I: 1st march 2011 to 3th april 2013 Phase II: 31th october 2014 to 1st june 2016.
  Recruitment took place in nine specialized treatment center in the province of Quebec (Canada).
Pre-assignment Details: Eighteen couples took part in the research eligibility, but they weren't enrolled in the study based on the exclusion criteria of the study :n=4 Low commitment towards relationship;n=4 Problematic alcohol/drug use [gambler]; n=3 Severe violence last 12 month; n=2 Low risk gambling [gambler]; n=2 Serious mental health problems [partner]; n=1 Partner with a gambling disorder ; n=1 Cohabitation less then six month ;n=1 Refused categorization
Period: 3 Months Post-admission
Arm/Group | Integrative Couple Treatment for Pathological Gambling (ICT-PG) | Usual Individual/Group Treatment
Started | 44 | 36
Completed | 41 (Couple modality: 1 couple refused and one gambler refused but his partner continued) | 30
Not Completed | 3 | 6
Not completed — Lost to Follow-up | 1 | 5
Not completed — Withdrawal by Subject | 2 | 1
Period: 9 Months Post-admission
Arm/Group | Integrative Couple Treatment for Pathological Gambling (ICT-PG) | Usual Individual/Group Treatment
Started | 41 | 30
Completed | 38 | 26 (26 couples completed + 1 individual (partner lost))
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 3 | 1
Not completed — Withdrawal by Subject | 0 | 3
Period: 18 Months Post-admission
Arm/Group | Integrative Couple Treatment for Pathological Gambling (ICT-PG) | Usual Individual/Group Treatment
Started | 38 | 26
Completed | 35 | 21
Not Completed | 3 | 5
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Integrative Couple Treatment for Pathological Gambling: Already described in the "Intervention Description" section
  Couple therapy: The experimental couple treatment is offered over 8 to 12 sessions of 90 minutes. The couple treatment called (Integrative Couple Treatment for Pathological Gambling - ICT-PG) is inspired by the "Alcohol Behavior Couple Therapy" from Epstein and McCrady, to which the team added diverse components to adjust to gamblers. During the sessions, the focus is on a) reducing/stopping gambling behaviors, b) helping the partner to stop behaviors facilitating gambling habits and rise the frequency of behaviors incompatible with gambling habits and c) improve marital components (communication, sharing positive moments, negotiation, mutual support).
- Usual Individual/Group Treatment: Well described in the Intervention section
  Usual individual/group treatment: The control group receive individual or group treatment as already offered by the specialized centers in addiction.Their partner can receive individual intervention if desired.
- Total: Total of all reporting groups
Arm/Group | Integrative Couple Treatment for Pathological Gambling | Usual Individual/Group Treatment | Total
Number analyzed (Participants) | 44 | 36 | 80
Age, Categorical [Count of Participants; unit: Participants]
  Gamblers: <=18 years | 0 | 0 | 0
  Gamblers: Between 18 and 65 years | 42 | 35 | 77
  Gamblers: >=65 years | 2 | 1 | 3
  Partners: <=18 years | 0 | 0 | 0
  Partners: Between 18 and 65 years | 41 | 34 | 75
  Partners: >=65 years | 3 | 2 | 5
Age, Continuous [Mean (Standard Deviation); unit: years]
  Gamblers | 42 (14) | 41 (12) | 42 (13)
  Partners | 42 (13) | 40 (14) | 41 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Gamblers: Female | 13 | 7 | 20
  Gamblers: Male | 31 | 29 | 60
  Partners: Female | 31 | 30 | 61
  Partners: Male | 13 | 6 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 44 | 36 | 80

OUTCOME MEASURES:

1. Primary Outcome: Gambling Symptom Assessment Scale (G-SAS)
Description: Outcome measure for Gamblers
  The G-SAS is a 12-item self-rated scale designed to assess gambling symptom severity and change during treatment.
  Each 12-item scale has a score ranging from 0 - 4 (adjective anchors for 0 and 4 vary for each item but "0 means no symptoms" and "4 means extreme symptoms").
  All items ask for an average symptom based on the past 7 days (average urge, frequency, duration and control,thoughts associated with gambling,time spent on gambling,anticipatory tension and/or excitement, emotional distress).
  The total score ranges from 0 to 48.
  A score between 8 and 20 is an indicator of low urges to gamble, between 21 and 30, moderate urges, between 31 and 40 severe urges and a score of over 40 reveals the presence of extreme urges in the player.
Time Frame: Admission, 3, 9 and 18 month post-admission (The first admission was March 2011 and the last admission will be June 2016)
Population: Analysis Population is based on all participants (n= 80 couples) enrolled in the study. Over the 18 months of follow-up, a slight attrition of participants can be observed, explaining the difference between the overall number of participants analyzed and the number of participants analyzed per row.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integrative Couple Treatment for Pathological Gambling (ICT-PG) | Usual Individual/Group Treatment
Number analyzed (Participants) | 44 | 36
score on a scale
  Admission | 18.52 (1.08) | 16.66 (1.20)
  3 months post-admission: number analyzed (Participants) | 41 | 30
  3 months post-admission | 6.85 (1.14) | 12.39 (1.31)
  9 months post-admission: number analyzed (Participants) | 38 | 26
  9 months post-admission | 4.30 (1.17) | 11.08 (1.44)
  18 months post-admission: number analyzed (Participants) | 35 | 22
  18 months post-admission | 4.01 (1.21) | 10.80 (1.53)

2. Primary Outcome: Frequency of the Most Problematic Game
Description: Outcome Measure for Gamblers
  Among 12 types of gambling activities, the highest frequency of gambling behaviors for the past 6 months (never = 0; every or almost every day=5). Maximum score is 5. The higher is the score, the higher is the frequency.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integrative Couple Treatment for Pathological Gambling (ICT-PG) | Usual Individual/Group Treatment
Number analyzed (Participants) | 44 | 36
score on a scale
  Admission | 3.66 (.15) | 3.56 (.16)
  3 months post-admission: number analyzed (Participants) | 41 | 30
  3 months post-admission | 2.14 (.19) | 2.20 (.20)
  9 months post-admission: number analyzed (Participants) | 38 | 26
  9 months post-admission | 1.68 (.21) | 2.37 (.22)
  18 months post-admission: number analyzed (Participants) | 35 | 22
  18 months post-admission | 2.17 (.20) | 2.73 (.24)

3. Primary Outcome: Detection of Gambling Problems and Services Need ("Détection et Besoin d'Aide en Regard du Jeu Excessif- DÉBA-Jeu")
Description: Outcome Measure for Gamblers
  The DEBA-Jeu is a very brief screening grid comprising eight Likert-type items in five points (never = 0, always = 4). The eight items form a scale where the total score varies between 0 and 32. The suggested breaking points are as follows: 0 to 1 = No problem gambling; 2 to 5 =Problem gambling ; 6 to 24 = High probability of problem gambling.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integrative Couple Treatment for Pathological Gambling (ICT-PG) | Usual Individual/Group Treatment
Number analyzed (Participants) | 44 | 36
score on a scale
  Admission | 19.41 (.88) | 20.45 (.97)
  3 months post-admission: number analyzed (Participants) | 41 | 30
  3 months post-admission | 6.29 (.90) | 7.90 (1.07)
  9 months post-admission: number analyzed (Participants) | 38 | 26
  9 months post-admission | 4.47 (.95) | 6.01 (1.14)
  18 months post-admission: number analyzed (Participants) | 35 | 22
  18 months post-admission | 4.47 (.98) | 6.26 (1.27)

4. Primary Outcome: Canadian Problem Gambling Index (CPGI)
Description: Outcome measure for Gamblers
  The Canadian Problem Gambling Index (CPGI) is a 9-item measure with a 4-point Likert-type scale (0 = Never, 3 = Almost always).It asks questions about an individual's gambling habits in the last three months from four categories:
  Gambling involvement; Problem gambling behaviour; Adverse Consequences; Correlates of problem gambling.
  Scores for the nine items are summed, and the results are interpreted as follows: 0 = non-problem ; 1-4 = low risk; 5-7 = moderate risk; 8 and + (maximum 27) = probable pathological player.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integrative Couple Treatment for Pathological Gambling (ICT-PG) | Usual Individual/Group Treatment
Number analyzed (Participants) | 44 | 36
score on a scale
  Admission | 14.85 (.74) | 15.68 (.82)
  3 months post-admission: number analyzed (Participants) | 41 | 30
  3 months post-admission | 5.86 (.77) | 6.97 (.89)
  9 months post-admission: number analyzed (Participants) | 38 | 26
  9 months post-admission | 3.98 (.80) | 5.31 (.97)
  18 months post-admission: number analyzed (Participants) | 35 | 22
  18 months post-admission | 4.26 (.83) | 4.91 (1.08)

5. Primary Outcome: Canadian Dollars Spent on Gambling
Description: Outcome measure for Gamblers
  Total Money spent in canadian dollars for all gambling activities during the last 3 months previous each research interview.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: canadian dollars
Groups:
- Integrative Couple Treatment for Pathological Gambling (ICT-PG): Couple therapy: The experimental couple treatment is offered over 8 to 12 sessions of 90 minutes. The couple treatment called (Integrative Couple Therapy for Pathological Gambling - ICT-PG) is inspired by the "Alcohol Behavior Couple Therapy" from Epstein and McCrady, to which the team added diverse components to adjust to gamblers. During the sessions, the focus is on a) reducing/stopping gambling behaviors, b) helping the partner to stop behaviors facilitating gambling habits and rise the frequency of behaviors incompatible with gambling habits and c) improve marital components (communication, sharing positive moments, negotiation, mutual support).
Arm/Group | Integrative Couple Treatment for Pathological Gambling (ICT-PG) | Usual Individual/Group Treatment
Number analyzed (Participants) | 44 | 36
canadian dollars
  Admission | 4587.87 (483.66) | 4244.70 (534.75)
  3 months post-admission: number analyzed (Participants) | 41 | 30
  3 months post-admission | 452.53 (500.54) | 825.71 (582.02)
  9 months post-admission: number analyzed (Participants) | 38 | 26
  9 months post-admission | 351.49 (517.16) | 390.14 (620.98)
  18 months post-admission: number analyzed (Participants) | 35 | 22
  18 months post-admission | 1062.09 (535.53) | 446.57 (681.53)

6. Primary Outcome: Impaired Control Over Gambling Scale (ICOG)
Description: Outcome Measure for Gamblers
  The ICOG is used to measure two aspects of control related to the JHA processes, namely the level of control over the desire to start playing (e.g., when I decide not to play, I watch stick to that decision) as well as the level of control once the game has started (e.g., when I knew I had little time to play, I would limit myself to the scheduled time). This questionnaire has a total of 10 items and uses a 5-point Likert-type scale ranging from "Never = 1" to "Always = 5", with 4 inverted items.
  The total score varies between 10 and 50. A high control represents a score between 10 and 16, a moderate control between 17 and 23 and a score of 24 and more presents a low control in the player.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integrative Couple Treatment for Pathological Gambling (ICT-PG) | Usual Individual/Group Treatment
Number analyzed (Participants) | 44 | 36
score on a scale
  Admission | 35.95 (1.29) | 37.92 (1.44)
  3 months post-admission: number analyzed (Participants) | 41 | 30
  3 months post-admission | 17.89 (1.34) | 22.31 (1.58)
  9 months post-admission: number analyzed (Participants) | 38 | 26
  9 months post-admission | 16.11 (1.41) | 20.59 (1.69)
  18 months post-admission: number analyzed (Participants) | 35 | 22
  18 months post-admission | 15.69 (1.45) | 18.26 (1.86)

7. Primary Outcome: Inventory of Erroneous Beliefs Related to Gambling ("Inventaire Des Croyances liées Aux Jeux" - ICROLJ)-Gambler
Description: Outcome Measure for Gamblers
  This questionnaire measures people's beliefs about gambling. The ICROLJ has 29 items and uses a 4-point Likert-type scale ranging from "Strongly disagree" = 0 to "Strongly agree"=4. To compute a total score, all item' score are summed. The total score ranges from 0 to 116.Higher the score is, more it indicates the presence of erroneous beliefs.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integrative Couple Treatment for Pathological Gambling (ICT-PG) | Usual Individual/Group Treatment
Number analyzed (Participants) | 44 | 36
score on a scale
  Admission | 52.67 (1.38) | 54.23 (1.53)
  3 months post-admission: number analyzed (Participants) | 41 | 30
  3 months post-admission | 39.44 (1.44) | 44.78 (1.67)
  9 months post-admission: number analyzed (Participants) | 38 | 26
  9 months post-admission | 39.11 (1.48) | 43.26 (1.79)
  18 months post-admission: number analyzed (Participants) | 35 | 22
  18 months post-admission | 38.90 (1.56) | 43.86 (1.94)

8. Primary Outcome: Negative Gambling Consequences-Gambler
Description: Outcome Measure for Gamblers
  Short questionnaire of 10 items, assessing to what extent the respondent considers his gambling habits in the last 6 months have harmed various aspects of his life (financial, living conditions, marital, physical health, professional life, social, legal and family). A 5-point Likert-type scale is used "Not at all = 0" to "Extremely = 4". To compute a total score, all item' score are summed. The total score ranges from 0 to 40.Higher the score is, more it's indicate that the respondent is experiencing negative impacts because of his gambling habits.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integrative Couple Treatment for Pathological Gambling (ICT-PG) | Usual Individual/Group Treatment
Number analyzed (Participants) | 44 | 36
score on a scale
  Admission | 16.83 (1.06) | 18.56 (1.17)
  3 months post-admission: number analyzed (Participants) | 41 | 30
  3 months post-admission | 6.84 (1.12) | 8.04 (1.30)
  9 months post-admission: number analyzed (Participants) | 38 | 26
  9 months post-admission | 4.96 (1.14) | 5.41 (1.38)
  18 months post-admission: number analyzed (Participants) | 35 | 22
  18 months post-admission | 4.40 (1.32) | 5.22 (1.61)

9. Primary Outcome: Negative Gambling Consequences-Partner
Description: Outcome Measure for Partners
  Short questionnaire of 10 items, assessing to what extent the respondent considers that his partner's gambling habits have harmed various aspects of his life in the last 6 months (financial, living conditions, marital, physical health, professional life, social, legal and family). A 5-point Likert-type scale is used "Not at all = 0" to "Extremely = 4". To compute a total score, all item' score are summed. The total score ranges from 0 to 40. Higher the score is, more it's indicate that the respondent is experiencing negative impacts because of his partner's gambling habits.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integrative Couple Treatment for Pathological Gambling (ICT-PG) | Usual Individual/Group Treatment
Number analyzed (Participants) | 44 | 36
score on a scale
  Admission | 17.65 (0.65) | 17.77 (0.72)
  3 months post-admission: number analyzed (Participants) | 41 | 30
  3 months post-admission | 8.57 (0.67) | 9.38 (0.76)
  9 months post-admission: number analyzed (Participants) | 38 | 26
  9 months post-admission | 5.30 (0.68) | 5.13 (0.79)
  18 months post-admission: number analyzed (Participants) | 35 | 22
  18 months post-admission | 5.89 (0.74) | 6.59 (0.89)

10. Primary Outcome: Inventory of Erroneous Beliefs Related to Gambling ("Inventaire Des Croyances liées Aux Jeux" - ICROLJ)-Partner
Description: Outcome Measure for Partners
  This questionnaire measures people's beliefs about gambling. The ICROLJ has 29 items and uses a 4-point Likert-type scale ranging from "Strongly disagree" = 0 to "Strongly agree"=4.
  To compute a total score, all item' score are summed. The total score ranges from 0 to 116. Higher the score is, more it indicates the presence of erroneous beliefs.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integrative Couple Treatment for Pathological Gambling (ICT-PG) | Usual Individual/Group Treatment
Number analyzed (Participants) | 44 | 36
score on a scale
  Admission | 40.74 (0.98) | 41.05 (1.08)
  3 months post-admission: number analyzed (Participants) | 41 | 30
  3 months post-admission | 35.03 (0.99) | 43.22 (1.12)
  9 months post-admission: number analyzed (Participants) | 38 | 26
  9 months post-admission | 37.12 (1.01) | 42.84 (1.13)
  18 months post-admission: number analyzed (Participants) | 35 | 22
  18 months post-admission | 37.38 (1.02) | 41.08 (1.19)

11. Secondary Outcome: Conjugal Support Questionnaire (CSQ)-Partner
Description: Outcome Measure for Partners
  This questionnaire measure the quality of the support received and given perceived by the two members of the couple. It consists of a total of 8 questions, with a 5-point Likert scale (1 = never; 5 = always).
  The total score shows support received and support gave, higher is the result, more it indicates that the member of the couple gave support and receives it (score min = 0 and score max=40).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integrative Couple Treatment for Pathological Gambling (ICT-PG) | Usual Individual/Group Treatment
Number analyzed (Participants) | 44 | 36
score on a scale
  Admission | 29.93 (0.46) | 29.90 (0.51)
  3 months post-admission: number analyzed (Participants) | 41 | 30
  3 months post-admission | 32.05 (0.47) | 29.46 (0.53)
  9 months post-admission: number analyzed (Participants) | 38 | 26
  9 months post-admission | 30.83 (0.47) | 31.09 (0.54)
  18 months post-admission: number analyzed (Participants) | 35 | 22
  18 months post-admission | 31.85 (0.49) | 30.99 (0.58)

12. Secondary Outcome: Psychological Distress Index (IDPESQ-14)-Partner
Description: Outcome Measure for Partners
  This instrument is used to measure psychological distress, including symptoms of depression and anxiety. We used the version of the questionnaire with 14 items. A Likert-type scale ranging from "never = 1" to "very often = 3" is used and the respondent must respond according to their condition during the last seven days. To compute a total score, all item' score are summed. The total score ranges from 0 to 42. A score of 26 and above indicates a high level of psychological distress.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integrative Couple Treatment for Pathological Gambling (ICT-PG) | Usual Individual/Group Treatment
Number analyzed (Participants) | 44 | 36
score on a scale
  Admission | 23.75 (.97) | 22.38 (1.08)
  3 months post-admission: number analyzed (Participants) | 41 | 30
  3 months post-admission | 12.76 (.99) | 16.4 (1.13)
  9 months post-admission: number analyzed (Participants) | 38 | 27
  9 months post-admission | 11.94 (1.01) | 17.03 (1.16)
  18 months post-admission: number analyzed (Participants) | 35 | 20
  18 months post-admission | 13.45 (1.04) | 16.96 (1.25)

13. Secondary Outcome: Center for Epidemiologic Studies Depression Scale (CES-D)-Partner
Description: Outcome Measure for Partners
  This instrument is used to measure depressive symptoms in an individual. It measures these symptoms as defined in the American Psychiatric Association Diagnostic and Statistical Manual (DSM-IV) for depressive episodes.This questionnaire has 20 items and it assesses how the psychological well-being of the person during the last week. A 4-point Likert-type scale is used ranging from "0 = Never, very rarely (less than a day)" to a rating of "3 = Frequently, all the time (5 to 7 days)" The score can therefore vary from 0 to 60, the higher it is the higher the risk of depression. For a man, a threshold of 17 indicates a risk of depression and for a woman the same threshold is 23.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integrative Couple Treatment for Pathological Gambling (ICT-PG) | Usual Individual/Group Treatment
Number analyzed (Participants) | 44 | 36
score on a scale
  Admission | 16.71 (.76) | 15.67 (.85)
  3 months post-admission: number analyzed (Participants) | 41 | 30
  3 months post-admission | 8.81 (.78) | 11.63 (.89)
  9 months post-admission: number analyzed (Participants) | 38 | 27
  9 months post-admission | 8.37 (.79) | 12.46 (.92)
  18 months post-admission: number analyzed (Participants) | 35 | 20
  18 months post-admission | 8.07 (.82) | 11.81 (.99)

14. Secondary Outcome: Psychological Distress Index (IDPESQ-14)-Gambler
Description: Outcome Measure for Gamblers
  This instrument is used to measure psychological distress, including symptoms of depression and anxiety. We used the version of the questionnaire with 14 items. A Likert-type scale ranging from "never = 1" to "very often = 3" is used and the respondent must respond according to their condition during the last seven days. To compute a total score, all item' score are summed. The total score ranges from 0 to 42. A score of 26 and above indicates a high level of psychological distress.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integrative Couple Treatment for Pathological Gambling (ICT-PG) | Usual Individual/Group Treatment
Number analyzed (Participants) | 44 | 36
score on a scale
  Admission | 18.83 (1.43) | 20.58 (1.58)
  3 months post-admission: number analyzed (Participants) | 41 | 30
  3 months post-admission | 14.45 (1.48) | 14.04 (1.73)
  9 months post-admission: number analyzed (Participants) | 38 | 26
  9 months post-admission | 10.19 (1.53) | 15.26 (1.84)
  18 months post-admission: number analyzed (Participants) | 35 | 22
  18 months post-admission | 12.24 (1.59) | 13.43 (2.04)

15. Secondary Outcome: Center for Epidemiologic Studies Depression Scale (CES-D)-Gambler
Description: Outcome Measure for Gamblers
  This instrument is used to measure depressive symptoms in an individual. It measures these symptoms as defined in the American Psychiatric Association Diagnostic and Statistical Manual (DSM-IV) for depressive episodes.This questionnaire has 20 items and it assesses how the psychological well-being of the person during the last week. A 4-point Likert-type scale is used ranging from "0 = Never, very rarely (less than a day)" to a rating of "3 = Frequently, all the time (5 to 7 days)" The score can therefore vary from 0 to 60, the higher it is the higher the risk of depression. For a man, a threshold of 17 indicates a risk of depression and for a woman the same threshold is 23.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integrative Couple Treatment for Pathological Gambling (ICT-PG) | Usual Individual/Group Treatment
Number analyzed (Participants) | 44 | 36
score on a scale
  Admission | 14.88 (1.03) | 15.56 (1.14)
  3 months post-admission: number analyzed (Participants) | 41 | 30
  3 months post-admission | 9.08 (1.06) | 11.86 (1.24)
  9 months post-admission: number analyzed (Participants) | 38 | 26
  9 months post-admission | 8.29 (1.10) | 10.96 (1.33)
  18: number analyzed (Participants) | 35 | 22
  18 | 9.01 (1.15) | 10.22 (1.48)

16. Secondary Outcome: Conjugal Support Questionnaire(CSQ)-Gambler
Description: Outcome Measure for Gamblers
  This questionnaire makes it possible to measure the quality of the support received and given perceived by the two members of the couple. It consists of a total of 8 questions, with a 5-point Likert scale (1 = never; 5 = always).
  The total score shows support received and support gave, higher is the result, more it indicates that the member of the couple gave support and receives it (score min = 0 and score max=40).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integrative Couple Treatment for Pathological Gambling (ICT-PG) | Usual Individual/Group Treatment
Number analyzed (Participants) | 44 | 36
score on a scale
  Admission | 31.10 (.46) | 30.68 (.51)
  3 months post-admission: number analyzed (Participants) | 41 | 30
  3 months post-admission | 32.65 (.48) | 30.77 (.56)
  9 months post-admission: number analyzed (Participants) | 38 | 26
  9 months post-admission | 33.30 (.49) | 30.64 (.59)
  18 months post-admission: number analyzed (Participants) | 35 | 22
  18 months post-admission | 33.67 (.54) | 29.66 (.67)

17. Secondary Outcome: Marital Status Inventory (MSI)-Partner
Description: Outcome Measure for Partners
  The MSI is used to measure marital stability in a couple. It comprises a series of 14 items (with inverted items) in a "true" or "false" format thus aiming to assess the risk of separation in this couple (e.g., I very often have ideas of divorce, until once a week or more). Marital distress is measured in terms of concrete actions taken by members of the couple in order to end their union. The total score is between 0 and 14. The higher the scores, the higher the risk of separation and marital distress. A threshold of 8 is considered to be a severe indicator of separation.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integrative Couple Treatment for Pathological Gambling (ICT-PG) | Usual Individual/Group Treatment
Number analyzed (Participants) | 44 | 36
score on a scale
  Admission | 4.14 (0.23) | 4.10 (0.26)
  3 months post-admission: number analyzed (Participants) | 41 | 30
  3 months post-admission | 2.19 (0.24) | 3.59 (0.27)
  9 months post-admission: number analyzed (Participants) | 38 | 26
  9 months post-admission | 2.26 (0.24) | 2.15 (0.28)
  18 months post-admission: number analyzed (Participants) | 35 | 22
  18 months post-admission | 2.17 (0.25) | 3.33 (0.31)

18. Secondary Outcome: Marital Status Inventory (MSI)-Gambler
Description: Outcome Measure for Gamblers
  The MSI is used to measure marital stability in a couple.
  It comprises a series of 14 items (with inverted items) in a "true" or "false" format thus aiming to assess the risk of separation in this couple (e.g., I very often have ideas of divorce, until once a week or more). Marital distress is measured in terms of concrete actions taken by members of the couple in order to end their union. The total score is between 0 and 14. The higher the scores, the higher the risk of separation and marital distress. A threshold of 8 is considered to be a severe indicator of separation.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integrative Couple Treatment for Pathological Gambling (ICT-PG) | Usual Individual/Group Treatment
Number analyzed (Participants) | 44 | 36
score on a scale
  Admission | 2.02 (0.25) | 2.18 (0.28)
  3 months post-admission: number analyzed (Participants) | 41 | 30
  3 months post-admission | 1.48 (0.26) | 1.91 (0.30)
  9 months post-admission: number analyzed (Participants) | 38 | 26
  9 months post-admission | 1.90 (0.27) | 1.65 (0.32)
  18 months post-admission: number analyzed (Participants) | 35 | 22
  18 months post-admission | 1.27 (.30) | 3.63 (.38)

19. Secondary Outcome: Dyadic Adjustment Scale (DAS-4)-Partner
Description: Outcome Measure for Partners
  The Dyadic Adjustment Scale is an ultra-brief measure degree of marital satisfaction within the couple.
  The short version is made up of only 4 items (considered divorce, estimation of the quality of the relation, confide to mate, degree of happiness): three of which are on a 6-point Likert scale ranging from 0 (all the time) to 5 (never) , while the final item is on a 7-point scale ranging from 0 (extremely happy) to 6 (perfect).
  Theoretically possible maximum score of 21, and minimum 0. Scores lower than 11 indicating relationship distress, scores between 12 and 14 corresponding to medium satisfaction and scores upper 15 indicating good marital satisfaction.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integrative Couple Treatment for Pathological Gambling (ICT-PG) | Usual Individual/Group Treatment
Number analyzed (Participants) | 44 | 36
score on a scale
  Admission | 11.67 (0.32) | 11.29 (0.35)
  3 months post-admission: number analyzed (Participants) | 41 | 30
  3 months post-admission | 15.42 (0.32) | 13.28 (0.37)
  9 months post-admission: number analyzed (Participants) | 38 | 26
  9 months post-admission | 15.35 (0.34) | 14.76 (0.38)
  18 months post-admission: number analyzed (Participants) | 35 | 22
  18 months post-admission | 15.05 (0.35) | 12.38 (0.41)

20. Secondary Outcome: Dyadic Adjustment Scale (DAS-4)-Gambler
Description: Outcome Measure for Gamblers
  The Dyadic Adjustment Scale is an ultra-brief measure degree of marital satisfaction within the couple.
  The short version is made up of only 4 items (considered divorce, estimation of the quality of the relation, confide to mate, degree of happiness): three of which are on a 6-point Likert scale ranging from 0 (all the time) to 5 (never) , while the final item is on a 7-point scale ranging from 0 (extremely happy) to 6 (perfect).
  Theoretically possible maximum score of 21, and minimum 0. Scores lower than 11 indicating relationship distress, scores between 12 and 14 corresponding to medium satisfaction and scores upper 15 indicating good marital satisfaction.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integrative Couple Treatment for Pathological Gambling (ICT-PG) | Usual Individual/Group Treatment
Number analyzed (Participants) | 44 | 36
score on a scale
  Admission | 11.96 (0.48) | 11.20 (0.53)
  3 months post-admission: number analyzed (Participants) | 41 | 30
  3 months post-admission | 15.09 (0.49) | 14.29 (0.58)
  9 months post-admission: number analyzed (Participants) | 38 | 26
  9 months post-admission | 16.08 (0.51) | 14.49 (0.61)
  18 months post-admission: number analyzed (Participants) | 35 | 22
  18 months post-admission | 15.43 (0.55) | 12.30 (0.70)

21. Secondary Outcome: Conflict Tactics Scale-2_Psychological Violence Issued by the Partner
Description: Outcome Measure for Gamblers
  The psychological violence suffered is a subscale of the CTS-2 questionnaire which aims to assess the manifestations of psychological violence committed against the Gambler in the last 3 months. It is made up of 14 items that are rated on a 7-point Likert scale (never happened = 0, 1 time = 1, 2 times = 2, 3 to 5 times = 3, 6 to 10 times = 4, 11 to 20 = 5, more than 20 times = 6). To compute a total score, all item' score are summed. The total score ranges from 0 to 84. The higher it is, more it indicates that the respondent has suffered episodes of violence.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integrative Couple Treatment for Pathological Gambling (ICT-PG) | Usual Individual/Group Treatment
Number analyzed (Participants) | 44 | 36
score on a scale
  Admission | 19.64 (1.78) | 19.17 (1.95)
  3 months post-admission: number analyzed (Participants) | 41 | 30
  3 months post-admission | 13.38 (1.84) | 14.16 (2.12)
  9 months post-admission: number analyzed (Participants) | 38 | 26
  9 months post-admission | 8.65 (1.94) | 12.46 (2.32)
  18 months post-admission: number analyzed (Participants) | 35 | 22
  18 months post-admission | 7.96 (2.05) | 14.52 (2.58)

22. Secondary Outcome: Interpersonal Communication Skills Inventory-self _Partner
Description: Outcome Measure for Partners
  This lists of skills consist of 17 items that expressed in statements representing observable verbal behaviors.Participants were asked to report frequency estimates of their own use of such verbal behaviors using a 4 point likert scale (0 = almost never, 4 = almost always). To compute a total score, all item' score are summed. The total score ranges from 0 to 68. The higher the score is, more it indicates the presence of good communication skills.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integrative Couple Treatment for Pathological Gambling (ICT-PG) | Usual Individual/Group Treatment
Number analyzed (Participants) | 44 | 36
score on a scale
  Admission | 37.39 (.53) | 36.99 (.58)
  3 months post-admission: number analyzed (Participants) | 41 | 30
  3 months post-admission | 38.69 (.54) | 38.45 (.61)
  9 months post-admission: number analyzed (Participants) | 38 | 27
  9 months post-admission | 39.73 (.54) | 38.42 (.62)
  18 months post-admission: number analyzed (Participants) | 35 | 20
  18 months post-admission | 39.82 (.57) | 39.24 (.67)

23. Secondary Outcome: Marital Problem Solving Scale (MPSS)-Gambler
Description: Outcome Measure for Gamblers
  This instrument has 9 items, using a 7-point Likert-type scale. It is used in order to better understand the negotiation and conflict resolution skills that the couple members have used within their marital relationship in the last three months.
  The score varies between 9 and 63. A high score indicates a greater degree of perceived problem-solving skill within the marital relationship.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integrative Couple Treatment for Pathological Gambling (ICT-PG) | Usual Individual/Group Treatment
Number analyzed (Participants) | 44 | 36
score on a scale
  Admission | 45.95 (.95) | 44.67 (1.05)
  3 months post-admission: number analyzed (Participants) | 41 | 30
  3 months post-admission | 48.53 (.98) | 46.63 (1.15)
  9 months post-admission: number analyzed (Participants) | 38 | 26
  9 months post-admission | 48.3 (1.02) | 44.75 (1.23)
  18 months post-admission: number analyzed (Participants) | 35 | 22
  18 months post-admission | 48.29 (1.12) | 44.7 (1.4)

24. Secondary Outcome: Coping Skills _Social Support Sub-scale_Gambler
Description: Outcome Measure for Gamblers
  This questionnaire is used to identify the coping strategies used to cope with gambling's habits in the last three months. The subscale is made up of 6 items marked from 0 to 3 (0 = not used; 3 = used a lot). To compute a total score, all item' score are summed. The total score ranges from 0 to 18. Higher the score is, more it indicates the respondent's tendency to adopt the behaviors described by the subscale when he is in a stressful situation.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integrative Couple Treatment for Pathological Gambling (ICT-PG) | Usual Individual/Group Treatment
Number analyzed (Participants) | 44 | 36
score on a scale
  Admission | 5.24 (.62) | 5.60 (.69)
  3 months post-admission: number analyzed (Participants) | 41 | 30
  3 months post-admission | 9.33 (.64) | 6.92 (.76)
  9 months post-admission: number analyzed (Participants) | 38 | 26
  9 months post-admission | 5.36 (.68) | 4.76 (.80)
  18 months post-admission: number analyzed (Participants) | 35 | 22
  18 months post-admission | 4.12 (.77) | 3.00 (.89)

25. Secondary Outcome: Standard Units of Alcoholic Drinks Per Week _Gambler
Description: Outcome measure for Gamblers
  Number of alcohol standard units (Canada, 1 unit = 13,6g of alcohol) per week during the last three months.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: standard units of alcoholic drinks
Arm/Group | Integrative Couple Treatment for Pathological Gambling (ICT-PG) | Usual Individual/Group Treatment
Number analyzed (Participants) | 44 | 36
standard units of alcoholic drinks
  Admission | 5.46 (1.10) | 4.96 (1.22)
  3 months post-admission: number analyzed (Participants) | 41 | 30
  3 months post-admission | 7.35 (1.14) | 4.15 (1.33)
  9 months post-admission: number analyzed (Participants) | 38 | 26
  9 months post-admission | 3.70 (1.18) | 4.28 (1.43)
  18 months post-admission: number analyzed (Participants) | 35 | 22
  18 months post-admission | 3.99 (1.25) | 7.47 (1.59)

26. Secondary Outcome: Frequency of Cannabis Use Per week_Gambler
Description: Outcome measure for Gamblers
  Frequency of cannabis use per week in the last three months with a 5-point Likert-type scale (never = 0, 3 times a week or more = 4). Higher the score is, more it indicates a high frequency of cannabis use.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integrative Couple Treatment for Pathological Gambling (ICT-PG) | Usual Individual/Group Treatment
Number analyzed (Participants) | 44 | 36
score on a scale
  Admission | .46 (.07) | .41 (.08)
  3 months post-admission: number analyzed (Participants) | 41 | 30
  3 months post-admission | .31 (.07) | .41 (.08)
  9 months post-admission: number analyzed (Participants) | 38 | 26
  9 months post-admission | .33 (.07) | .41 (.09)
  18 months post-admission: number analyzed (Participants) | 35 | 22
  18 months post-admission | .36 (.08) | .54 (.09)

27. Secondary Outcome: Conflict Tactics Scale-2 _ Physical Violence Issued by the Partner
Description: Outcome measure for Gamblers
  The physical violence suffered is a subscale of the CTS-2 questionnaire which aims to assess the manifestations of physical violence committed against the Gambler in the last 3 months. It is made up of 18 items that are rated on a 7-point Likert scale (never happened = 0, 1 time = 1, 2 times = 2, 3 to 5 times = 3, 6 to 10 times = 4, 11 to 20 = 5, more than 20 times = 6). The total score corresponds to the average obtained on the 18 items, the higher it is, more it indicates that the respondent has suffered episodes of violence.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integrative Couple Treatment for Pathological Gambling (ICT-PG) | Usual Individual/Group Treatment
Number analyzed (Participants) | 44 | 36
score on a scale
  Admission | 0.47 (.49) | 1.21 (.42)
  3 months post-admission: number analyzed (Participants) | 41 | 30
  3 months post-admission | 0.82 (.42) | 1.34 (.38)
  9 months post-admission: number analyzed (Participants) | 38 | 26
  9 months post-admission | .87 (.56) | 1.55 (.46)
  18 months post-admission: number analyzed (Participants) | 35 | 22
  18 months post-admission | .38 (.45) | 1.68 (.40)

28. Secondary Outcome: Conflict Tactics Scale-2_ Physique Violence Issued by the Gambler
Description: Outcome Measure for the Partner
  The physical violence suffered is a subscale of the CTS-2 questionnaire which aims to assess the manifestations of physical violence committed against the partner in the last 3 months. It is made up of 18 items that are rated on a 7-point Likert scale (never happened = 0, 1 time = 1, 2 times = 2, 3 to 5 times = 3, 6 to 10 times = 4, 11 to 20 = 5, more than 20 times = 6). The total score corresponds to the average obtained on the 18 items, the higher it is, more it indicates that the respondent has suffered episodes of violence.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integrative Couple Treatment for Pathological Gambling (ICT-PG) | Usual Individual/Group Treatment
Number analyzed (Participants) | 44 | 36
score on a scale
  Admission | 1.42 (.31) | 1.69 (.35)
  3 months post-admission: number analyzed (Participants) | 41 | 30
  3 months post-admission | 1.23 (.32) | 1.71 (.36)
  9 months post-admission: number analyzed (Participants) | 38 | 27
  9 months post-admission | .94 (.32) | .79 (.38)
  18 months post-admission: number analyzed (Participants) | 35 | 20
  18 months post-admission | .46 (.34) | 1.56 (.40)

29. Secondary Outcome: Conflict Tactics Scale-2 _ Psychological Violence Issued by the Gambler
Description: Outcome Measure for Partners
  The psychological violence suffered is a subscale of the CTS-2 questionnaire which aims to assess the manifestations of psychological violence committed against the partner in the last 3 months. It is made up of 14 items that are rated on a 7-point Likert scale (never happened = 0, 1 time = 1, 2 times = 2, 3 to 5 times = 3, 6 to 10 times = 4, 11 to 20 = 5, more than 20 times = 6). To compute a total score, all item' score are summed. The total score ranges from 0 to 84. The higher it is, more it indicates that the respondent has suffered episodes of violence.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integrative Couple Treatment for Pathological Gambling (ICT-PG) | Usual Individual/Group Treatment
Number analyzed (Participants) | 44 | 36
score on a scale
  Admission | 21.50 (1.40) | 23.44 (1.53)
  3 months post-admission: number analyzed (Participants) | 41 | 30
  3 months post-admission | 17.44 (1.43) | 18.36 (1.61)
  9 months post-admission: number analyzed (Participants) | 38 | 27
  9 months post-admission | 14.91 (1.46) | 16.52 (1.66)
  18 months post-admission: number analyzed (Participants) | 20 | 35
  18 months post-admission | 11.09 (1.54) | 17.00 (1.81)

30. Secondary Outcome: Coping Skills _Positive Reevaluation/Problem Solving Sub-scale_Gambler
Description: Outcome measure for Gamblers
  This questionnaire is used to identify the coping strategies used to cope with gambling's habits in the last three months. The subscale is made up of 9 items marked from 0 to 3 (0 = not used; 3 = used a lot). To compute a total score, all item' score are summed. The total score ranges from 0 to 27. Higher the score is, more it indicates the respondent's tendency to adopt the behaviors described by the subscale when he is in a stressful situation.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Couple Treatment for Pathological Gambling: Already described in the "Intervention Description" section
  Couple therapy: The experimental couple treatment is offered over 8 to 12 sessions of 90 minutes. The couple treatment called (Integrative Couple Treatment for Pathological Gambling - ICT-PG) is inspired by the "Alcohol Behavior Couple Therapy" from Epstein and McCrady, to which the team added diverse components to adjust to gamblers. During the sessions, the focus is on a) reducing/stopping gambling behaviors, b) helping the partner to stop behaviors facilitating gambling habits and rise the frequency of behaviors incompatible with gambling habits and c) improve marital components (communication, sharing positive moments, negotiation, mutual support).
Arm/Group | Couple Treatment for Pathological Gambling | Usual Individual/Group Treatment
Number analyzed (Participants) | 44 | 36
score on a scale
  Admission | 10.08 (1.08) | 9.90 (1.21)
  3 months post-admission: number analyzed (Participants) | 41 | 30
  3 months post-admission | 15.48 (1.12) | 13.12 (1.33)
  9 months post-admission: number analyzed (Participants) | 38 | 26
  9 months post-admission | 10.69 (1.19) | 10.79 (1.40)
  18 months post-admission: number analyzed (Participants) | 35 | 22
  18 months post-admission | 9.25 (1.34) | 8.52 (1.55)

31. Secondary Outcome: Coping Skills _Distancing / Withdrawal Sub-scale_Gambler
Description: Outcome measure for Gamblers
  This questionnaire is used to identify the coping strategies used to cope with gambling's habits in the last three months. The subscale is made up of 6 items marked from 0 to 3 (0 = not used; 3 = used a lot). To compute a total score, all item' score are summed. The total score ranges from 0 to 18.Higher the score is, more it indicates the respondent's tendency to adopt the behaviors described by the subscale when he is in a stressful situation.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Couple Treatment for Pathological Gambling | Usual Individual/Group Treatment
Number analyzed (Participants) | 44 | 36
score on a scale
  Admission | 8.14 (.48) | 9.22 (.54)
  3 months post-admission: number analyzed (Participants) | 41 | 30
  3 months post-admission | 4.85 (.50) | 5.3 (.59)
  9 months post-admission: number analyzed (Participants) | 38 | 26
  9 months post-admission | 2.78 (.53) | 4.72 (.62)
  18 months post-admission: number analyzed (Participants) | 35 | 22
  18 months post-admission | 2.11 (.6) | 2.49 (.69)

32. Secondary Outcome: Marital Problem Solving Scale (MPSS)-Partner
Description: Outcome Measure for Partners This instrument has 9 items, using a 7-point Likert-type scale. It is used in order to better understand the negotiation and conflict resolution skills that the couple members have used within their marital relationship in the last three months.The score varies between 9 and 63. A high score indicates a greater degree of perceived problem-solving skill within the marital relationship.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integrative Couple Treatment for Pathological Gambling (ICT-PG) | Usual Individual/Group Treatment
Number analyzed (Participants) | 44 | 36
score on a scale
  Admission | 44.14 (.67) | 43.53 (.74)
  3 months post-admission: number analyzed (Participants) | 41 | 30
  3 months post-admission | 48.58 (.68) | 47.02 (.77)
  9 months post-admission: number analyzed (Participants) | 38 | 27
  9 months post-admission | 47.9 (.69) | 48.62 (.8)
  18 months post-admission: number analyzed (Participants) | 35 | 20
  18 months post-admission | 48.75 (.73) | 48.54 (.88)

33. Secondary Outcome: Interpersonal Communication Skills Inventory-self _Gambler
Description: Outcome Measure for Gamblers
  This lists of skills consist of 17 items that expressed in statements representing observable verbal behaviors.Participants were asked to report frequency estimates of their own use of such verbal behaviors using a 4 point likert scale (0 = almost never, 4 = almost always). To compute a total score, all item' score are summed. The total score ranges from 0 to 68.The higher the score is, more it indicates the presence of good communication skills.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integrative Couple Treatment for Pathological Gambling (ICT-PG) | Usual Individual/Group Treatment
Number analyzed (Participants) | 44 | 36
score on a scale
  Admission | 34.34 (.9) | 33.48 (1.00)
  3 months post-admission: number analyzed (Participants) | 41 | 30
  3 months post-admission | 38.57 (.94) | 34.48 (1.09)
  9 months post-admission: number analyzed (Participants) | 38 | 26
  9 months post-admission | 37.41 (.97) | 35.66 (1.17)
  18 months post-admission: number analyzed (Participants) | 35 | 22
  18 months post-admission | 39.68 (1.06) | 35.86 (1.32)

34. Secondary Outcome: Coping Skills _Social Support Sub-scale_Partner
Description: Outcome Measure for Partners
  This questionnaire is used to identify coping strategies to cope with stressful situations caused by their spouse's gambling habits in the last three months. The subscale is made up of 6 items marked from 0 to 3 (0 = not used; 3 = used a lot). To compute a total score, all item' score are summed. The total score ranges from 0 to 18.Higher the score is, more it indicates the respondent's tendency to adopt the behaviors described by the subscale when he is in a stressful situation.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integrative Couple Treatment for Pathological Gambling | Usual Individual/Group Treatment
Number analyzed (Participants) | 44 | 36
score on a scale
  Admission | 8.54 (0.61) | 8.50 (0.67)
  3 months post-admission: number analyzed (Participants) | 41 | 30
  3 months post-admission | 8.71 (0.62) | 6.02 (0.70)
  9 months post-admission: number analyzed (Participants) | 38 | 26
  9 months post-admission | 6.40 (0.63) | 5.63 (0.71)
  18 months post-admission: number analyzed (Participants) | 35 | 22
  18 months post-admission | 7.10 (0.70) | 8.11 (0.80)

35. Secondary Outcome: Coping Skills _Distancing / Withdrawal Sub-scale_Partner
Description: as for outcome 34
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Couple Treatment for Pathological Gambling | Usual Individual/Group Treatment
Number analyzed (Participants) | 44 | 36
score on a scale
  Admission | 5.38 (0.31) | 5.69 (0.34)
  3 months post-admission: number analyzed (Participants) | 41 | 30
  3 months post-admission | 2.95 (0.32) | 3.30 (0.36)
  9 months post-admission: number analyzed (Participants) | 38 | 26
  9 months post-admission | 2.50 (0.32) | 3.39 (0.36)
  18 months post-admission: number analyzed (Participants) | 35 | 22
  18 months post-admission | 2.48 (0.36) | 3.30 (0.42)

36. Secondary Outcome: Coping Skills_Positive Reevaluation/Problem Solving Sub-scale_Partner
Description: Outcome Measure for Partners
  This questionnaire is used to identify coping strategies to cope with stressful situations caused by their spouse's gambling habits in the last three months. The subscale is made up of 9 items marked from 0 to 3 (0 = not used; 3 = used a lot). To compute a total score, all item' score are summed. The total score ranges from 0 to 27.Higher the score is, more it indicates the respondent's tendency to adopt the behaviors described by the subscale when he is in a stressful situation.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Couple Treatment for Pathological Gambling | Usual Individual/Group Treatment
Number analyzed (Participants) | 44 | 36
score on a scale
  Admission | 8.54 (0.61) | 8.50 (0.67)
  3 months post-admission: number analyzed (Participants) | 41 | 30
  3 months post-admission | 8.71 (0.62) | 6.02 (0.70)
  9 months post-admission: number analyzed (Participants) | 38 | 26
  9 months post-admission | 6.40 (0.63) | 5.63 (0.71)
  18 months post-admission: number analyzed (Participants) | 35 | 22
  18 months post-admission | 7.10 (0.70) | 8.11 (0.80)

37. Secondary Outcome: Standard Units of Alcoholic Drinks Per Week _Partner
Description: Outcome measure for Partners
  Number of alcohol standard units (Canada, 1 unit = 13,6g of alcohol) per week during the last three months.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: standard units of alcoholic drinks
Arm/Group | Integrative Couple Treatment for Pathological Gambling (ICT-PG) | Usual Individual/Group Treatment
Number analyzed (Participants) | 44 | 36
standard units of alcoholic drinks
  Admission | 4.04 (0.40) | 3.89 (0.44)
  3 months post-admission: number analyzed (Participants) | 41 | 30
  3 months post-admission | 3.98 (0.40) | 3.87 (0.45)
  9 months post-admission: number analyzed (Participants) | 38 | 26
  9 months post-admission | 4.08 (0.41) | 3.69 (0.46)
  18 months post-admission: number analyzed (Participants) | 35 | 22
  18 months post-admission | 3.40 (0.42) | 3.47 (0.49)

38. Secondary Outcome: Frequency of Cannabis Use Per week_Partner
Description: Outcome measure for Partners
  Frequency of cannabis use per week in the last three months with a 5-point Likert-type scale (never = 0, 3 times a week or more = 4). Higher the score is, more it indicates a high frequency of cannabis use.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integrative Couple Treatment for Pathological Gambling (ICT-PG) | Usual Individual/Group Treatment
Number analyzed (Participants) | 44 | 36
score on a scale
  Admission | 0.24 (0.05) | 0.22 (0.06)
  3 months post-admission: number analyzed (Participants) | 41 | 30
  3 months post-admission | 0.29 (0.05) | 0.32 (0.06)
  9 months post-admission: number analyzed (Participants) | 38 | 26
  9 months post-admission | 0.21 (0.06) | 0.29 (0.06)
  18 months post-admission: number analyzed (Participants) | 35 | 22
  18 months post-admission | 0.21 (0.06) | 0.35 (0.07)

ADVERSE EVENTS:
Time Frame: We did not collect information on adverse events.
Description: Since our intervention was behavioral in nature and did not involve any biomedical follow-up, we had no data to report in this section.
Arm/Group | Integrative Couple Treatment for Pathological Gambling (ICT-PG) | Usual Individual/Group Treatment
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2015-02-15): https://cdn.clinicaltrials.gov/large-docs/85/NCT02240485/Prot_000.pdf
  • Statistical Analysis Plan (2015-02-15): https://cdn.clinicaltrials.gov/large-docs/85/NCT02240485/SAP_001.pdf
  • Informed Consent Form (2015-02-15): https://cdn.clinicaltrials.gov/large-docs/85/NCT02240485/ICF_002.pdf